CLINICAL TRIAL: NCT02102581
Title: Evaluation of Short-term Effects of Tourniquet Use in Different Ways During Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Evaluation of Short-term Effects of Tourniquet Use in Different Ways During Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Orthopedic deparment
Record Dates: First submitted 2014-03-24; First posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis
Keywords: Tourniquet; Total knee arthroplasty; Blood loss; Limb swelling; Limb circumference
MeSH Terms: conditions — Osteoarthritis; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- short time tourniquet: 60 patients were randomly divided into 2 groups (30 cases/group): group A using the tourniquet throughout the operation, and group B using the tourniquet starting from the implantation of prosthesis to the completion of the operation(short time).
  Interventions: Procedure: short time tourniquet

INTERVENTIONS:
Procedure: short time tourniquet — short time tourniquet: the tourniquet starting from the implantation of prosthesis to the completion of the operation.

SUMMARY:
To study the short-term effects of tourniquet use in different ways in total knee arthroplasty,60 patients were randomly divided into 2 groups (30 cases/group): group A using the tourniquet throughout the operation, and group B using the tourniquet starting from the implantation of prosthesis to the completion of the operation. Operation time, total measured blood loss, intraoperative transfusion volume, and complication were recorded. Hemoglobin level was recorded preoperatively and in postoperative 1, 3, 7 and 14 days, and the limb circumference, pain score, and knee joint range of motion were also recorded preoperatively and in postoperative 3,7 and 14 days.Investigators want to observe the difference between the two groups. Hypothesis was made that patients in group B may feel better after operation for short time use of tourniquet.

DETAILED DESCRIPTION:
Objective: To study the short-term effects of tourniquet use in different ways in total knee arthroplasty.

Methods: 60 patients were randomly divided into 2 groups (30 cases/group): group A using the tourniquet throughout the operation, and group B using the tourniquet starting from the implantation of prosthesis to the completion of the operation. Operation time, total measured blood loss, intraoperative transfusion volume, and complication were recorded. Hemoglobin level was recorded preoperatively and in postoperative 1, 3, 7 and 14 days, and the limb circumference, pain score, and knee joint range of motion were also recorded preoperatively and in postoperative 3,7 and 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the study included those who underwent initial unilateral TKA for osteoarthritis or rheumatoid arthritis.

Exclusion Criteria:

* Patients with diabetes, hemorrhagic disease, Hb < 100 g/L, peripheral neurovascular disease, malignant tumors, history of vascular thrombosis, or history of infection in the lower limb were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 consecutive patients who underwent routine TKA were included in this prospective randomized study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
the limb circumference at 10 cm above the knee at postoperative day 1,3,7 and 14 | 14 days after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yu Fan, MD, Principal Investigator — an orthopaedist of Peing Union Medical College Hospital
Locations (1):
- orthopedic department, Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Fan Y, Jin J, Sun Z, Li W, Lin J, Weng X, Qiu G. The limited use of a tourniquet during total knee arthroplasty: a randomized controlled trial. Knee. 2014 Dec;21(6):1263-8. doi: 10.1016/j.knee.2014.08.002. Epub 2014 Sep 9. PMID 25212990